CLINICAL TRIAL: NCT07269132
Title: Applying the ADDIE Model to Develop a Multimedia Educational Program to Enhance Chemotherapy Knowledge and Self-Efficacy Among ICU Nurses in a Medical Center in Southern Taiwan
Brief Title: Applying the ADDIE Model to Develop a Multimedia Program to Enhance Chemotherapy Knowledge and Self-Efficacy Among Intensive Care Unit Nurses
Acronym: ADDIE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A-ER-114-399
Record Dates: First submitted 2025-11-19; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Nurse; Self-Efficacy; eLearning; Chemotherapy; ICU
Keywords: ADDIE model; Interactive multimedia education; Chemotherapy nursing competence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Group Interactive Multimedia Learning Intervention (Experimental): Participants in this arm will receive access to an interactive multimedia learning system developed based on the ADDIE model (Analysis, Design, Development & Implementation, Evaluation). The system provides scenario-based modules covering chemotherapy drug administration procedures, error prevention, and adverse effect monitoring.
  Each participant will complete a pretest assessing baseline knowledge and self-efficacy, followed by a self-paced learning session using the multimedia system for approximately 30 minutes. After completing the learning activities, participants will take a posttest evaluating knowledge acquisition, changes in self-efficacy, and system usability using the System Usability Scale (SUS).
  This single-group intervention aims to enhance ICU nurses' competence, confidence, and learning engagement in chemotherapy care through an interactive, technology-enhanced educational approach.
  Interventions: Other: Interactive multimedia education

INTERVENTIONS:
Other: Interactive multimedia education — This intervention involves the implementation and evaluation of an interactive multimedia learning system developed to enhance nurses' competence and self-efficacy in chemotherapy administration. The system integrates clinical guidelines, audiovisual demonstrations, and scenario-based simulations designed according to the ADDIE instructional design model (Analysis, Design, Development & Implementation, Evaluation).
  Participants will first complete a pretest assessing baseline knowledge and self-efficacy, then independently access the multimedia learning platform to engage with modules covering chemotherapy drug administration procedures, error management, and adverse effect monitoring. The platform allows self-paced learning and provides instant feedback through interactive exercises. After completion, participants will take a posttest evaluating knowledge gain, self-efficacy improvement, and system usability.

SUMMARY:
Research Methods, Procedures, and Participant Requirements:

This study will test a multimedia interactive learning system designed to help nurses conveniently learn about chemotherapy drug administration. The study is scheduled to be conducted from November to December, 2025. Participants are expected to cooperate with the following procedures:

Pre-test: Complete a questionnaire that includes basic demographic information and a self-efficacy scale. The estimated time for completion is about 10 minutes.

System Experience: Use the multimedia learning system developed by the research team to study topics such as chemotherapy administration procedures, common error management, and side effect monitoring. The total learning time is approximately 30 minutes, and participants may use the system at their own pace-continuous use in one session is not required.

Post-test: After completing the learning session, participants will fill out another questionnaire assessing learning outcomes, changes in self-efficacy, user experience, and system usability. This takes approximately 15-20 minutes.

The total participation time is estimated to be 45-60 minutes. All responses will be collected anonymously. Participants may contact the research team at any time if they have questions or concerns, and assistance will be provided as needed.

DETAILED DESCRIPTION:
This study adopted a quasi-experimental research design using a one-group pretest-posttest approach, and participants were recruited through convenience sampling. The overall research framework followed the ADDIE model, which consists of four main phases: Analysis, Design, Development & Implementation, and Evaluation. The study integrated the clinical needs of the intensive care unit (ICU) to develop and apply an interactive multimedia educational program. The research process is described as follows:

1. Analysis Phase

   In this phase, the research team conducted a situational analysis in the ICU through on-site interviews and structured interview guides with nurses to gain a comprehensive understanding of the challenges they face during chemotherapy administration. The key areas of investigation included nurses' familiarity with drug characteristics, mastery of administration and standard procedures, monitoring of chemotherapy-related side effects, and their ability to respond to unexpected situations.

   To assess nurses' self-efficacy comprehensively, a self-efficacy questionnaire was distributed to collect data on their confidence and practical needs regarding chemotherapy administration and medication safety. The findings from this phase served as the foundation for the subsequent system design, ensuring that the system functions aligned closely with clinical practice needs.
2. Design Phase

   Based on the results of the analysis phase, the second phase focused on constructing a blueprint for the interactive multimedia education program. The research unit established an Oncology Treatment Task Force in 2021 and released a revised version of the "Oncology Treatment Manual" in the same year. The 32-page manual covers topics such as pre-administration assessment, introduction to common oral and injectable chemotherapy drugs, principles for handling medical orders, and procedures for managing extravasation. It also integrates audiovisual teaching resources to provide multiple learning channels.

   Drawing upon the manual and clinical requirements, the research team developed a scenario-based interactive multimedia design emphasizing common clinical issues and medication processes. This allows nurses to receive accurate, real-time guidance when encountering problems or seeking information in clinical practice.
3. Development & Implementation Phase

   In this phase, the research team developed and implemented the multimedia educational content and system interface based on the needs and materials identified in the previous stages. The process included functional development, content verification, and multiple rounds of pilot testing. ICU nurses were invited to test the system and provide feedback. The research team continuously refined the interface and content presentation according to user feedback to ensure that the educational system met real clinical requirements and was user-friendly.
4. Evaluation Phase

During the evaluation phase, the research team collected nurses' feedback after using the multimedia system. The evaluation incorporated the Technology Acceptance Model (TAM) and the System Usability Scale (SUS) to assess the system's usability and acceptance. If the results indicated areas for improvement, the team would return to the design or development phase for revision and optimization, achieving continuous iteration and quality enhancement of the system.

ELIGIBILITY:
The study site is located in the intensive care unit (ICU) of a medical center in southern Taiwan, and the primary participants are nurses working in this unit. Considering the characteristics of ICU work and its unique clinical environment, participating nurses are required to have sufficient clinical experience to ensure meaningful feedback and accurately reflect the practical impact of the interactive multimedia education program in real clinical settings.

Inclusion Criteria

* Participants must meet all of the following criteria:
* Currently employed as nurses in the Intensive Care Unit (ICU) and actively engaged in patient care involving chemotherapy ad-ministration or chemotherapy-related nursing responsibilities.

This ensures that participants possess foundational knowledge and clinical experience relevant to chemotherapy procedures.

Exclusion Criteria

* Participants meeting any of the following conditions will be excluded:
* Nurses who are temporarily away from clinical duties, such as those on personal leave, leave of absence, or unpaid leave.
* Nurses who are unable to participate consistently due to job reassignment or changes in work responsibilities.
* Nurses currently participating in other chemotherapy-related research that may interfere with data collection or study outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome (1) change in chemotherapy-related knowledge | Baseline (pretest) and immediately after completion of the multimedia learning intervention (posttest, approximately within 1 hour).
  Change in Knowledge
  Knowledge will be assessed using a structured questionnaire derived from the Oncology Treatment Manual, covering medication preparation, administration procedures, and the management of adverse effects. Objective knowledge will be measured using a 20-30 item multiple-choice exam based on the same content areas, with scores reported as percentage correct and pass rate (threshold ≥80%). Changes in knowledge scores from pretest to posttest will be used to evaluate the effect of the intervention.The score ranges from 0 to 100, with higher scores indicating better performance.
Self-Efficacy | Baseline (pretest) and immediately after completion of the multimedia learning intervention (posttest, approximately within 1 hour).
  Self-efficacy will be measured using the 10-item General Self-Efficacy Scale (GSES), a validated instrument assessing participants' confidence in safely performing chemotherapy-related nursing tasks. The scale is rated on a 4-point Likert format (score range: 10-40), with higher scores indicating stronger self-efficacy. Changes in self-efficacy scores from pretest to posttest will be used to determine the effect of the multimedia learning system. In this study, the GSES demonstrated high reliability (Cronbach's α = 0.940).

SECONDARY OUTCOMES:
System Usability | Immediately after completion of the multimedia learning intervention (within 1 hour).
  System usability was evaluated using the validated 10-item System Usability Scale (SUS), a widely applied instrument for assessing ease of use, interface quality, and overall user satisfaction. Items are rated on a five-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). SUS scoring follows the standard method: odd-numbered items are scored as response - 1, and even-numbered items as 5 - response, producing item scores from 0 to 4. The total score is then multiplied by 2.5 to yield a final SUS score ranging from 0 to 100, with higher scores indicating better usability. Scores ≥70 are generally considered acceptable, with higher thresholds reflecting good to excellent usability.
Technology Acceptance | Immediately after completion of the multimedia learning intervention (within 1 hour)
  System acceptance was assessed using an adapted 11-item Technology Acceptance Model (TAM) questionnaire covering perceived usefulness (PU), perceived ease of use (PEOU), and user attitude (UA). Items were rated on a five-point Likert scale (1 = strongly disagree, 5 = strongly agree), with higher scores indicating greater agreement. Domain scores were calculated as the mean of items within each construct. A total score (range: 11-55) was also derived by summing all items, with higher values indicating stronger overall system acceptance.

OTHER OUTCOMES:
Demographic variables | 3~5 minutes
  1. Gender: male or female.
  2. Clinical Professional Advancement Level: 01. N; 02. N1; 03. N2; 04. N3; 05. N4.
  3. Education Level: 01. Junior College; 02. Bachelor's Degree; 03. Master's Degree; 04. Doctoral Degree
  4. Total Nursing Work Experience:___ years ___ months
  5. Prior Work Experience in a Chemotherapy Ward Before Entering MICU (total years may be accumulated):___ years ___ months
Questionnaire | 3~5 minutes
  Have you handled antineoplastic (chemotherapy) drugs within the past month?Including verifying chemotherapy prescriptions or administering oral/injectable chemotherapy.01. Yes; 02. No

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsang SK, Hui EK, Law BC. Self-efficacy as a positive youth development construct: a conceptual review. ScientificWorldJournal. 2012;2012:452327. doi: 10.1100/2012/452327. Epub 2012 Apr 29. PMID 22645423
- [Background] Torous J, Chan SR, Yee-Marie Tan S, Behrens J, Mathew I, Conrad EJ, Hinton L, Yellowlees P, Keshavan M. Patient Smartphone Ownership and Interest in Mobile Apps to Monitor Symptoms of Mental Health Conditions: A Survey in Four Geographically Distinct Psychiatric Clinics. JMIR Ment Health. 2014 Dec 23;1(1):e5. doi: 10.2196/mental.4004. eCollection 2014 Jul-Dec. PMID 26543905
- [Background] Rosenberg, M. J. (2001). E-learning: Strategies for Delivering Knowledge in the Digital. Mcgraw- 2001.
- [Background] Morrison, G. R., Ross, S. J., Morrison, J. R., & Kalman, H. K. (2019). Designing effective instruction. John Wiley & Sons.
- [Background] Molenda, M. (2003). In search of the elusive ADDIE model. Performance improvement, 42(5), 34-37.
- [Background] McKimm J, Jollie C, Cantillon P. ABC of learning and teaching: Web based learning. BMJ. 2003 Apr 19;326(7394):870-3. doi: 10.1136/bmj.326.7394.870. No abstract available. PMID 12702625
- [Background] McCarthy BC Jr, Tuiskula KA, Driscoll TP, Davis AM. Medication errors resulting in harm: Using chargemaster data to determine association with cost of hospitalization and length of stay. Am J Health Syst Pharm. 2017 Dec 1;74(23 Supplement 4):S102-S107. doi: 10.2146/ajhp160848. PMID 29167147
- [Background] Klasnja P, Pratt W. Healthcare in the pocket: mapping the space of mobile-phone health interventions. J Biomed Inform. 2012 Feb;45(1):184-98. doi: 10.1016/j.jbi.2011.08.017. Epub 2011 Sep 9. PMID 21925288
- [Background] World Health Organization. (2017). Global diffusion of eHealth: making universal health coverage achievable: report of the third global survey on eHealth. World Health Organization.
- [Background] Bandura, A. (1997). Self-efficacy: The exercise of control. Macmillan.
- [Background] Bandura, A. (1986). Social foundations of thought and action. Englewood Cliffs, NJ, 1986 (23-28), 2.
- [Background] McCutcheon K, Lohan M, Traynor M, Martin D. A systematic review evaluating the impact of online or blended learning vs. face-to-face learning of clinical skills in undergraduate nurse education. J Adv Nurs. 2015 Feb;71(2):255-70. doi: 10.1111/jan.12509. Epub 2014 Aug 19. PMID 25134985
- [Background] Button D, Harrington A, Belan I. E-learning & information communication technology (ICT) in nursing education: A review of the literature. Nurse Educ Today. 2014 Oct;34(10):1311-23. doi: 10.1016/j.nedt.2013.05.002. Epub 2013 Jun 18. PMID 23786869